CLINICAL TRIAL: NCT02808286
Title: An Randomized Controlled Trial (RCT) Testing the Effectiveness of a Hybrid Emotion-focused Treatment for Chronic Pain Patients With Co-occurring Emotional Problems
Brief Title: A Hybrid Emotion-focused Treatment for Chronic Pain Patients With Emotional Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYBRID
Record Dates: First submitted 2016-06-01; First posted 2016-06-21 (Estimated); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hybrid (Experimental): The hybrid emotion-focused treatment consists of 10-15 individual 1/1,5 hour sessions. It includes the following stages (examples of methods in parathesis)
  Stage I. Analysis of emotions and pain (Validation, Compassion, Chain analysis, Values & goals).
  Stage II. Developing skills (Dialectics, Self-validation, Self-compassion, emotion regulation skills).
  Stage III. Exposure training (Exposure for emotionally sensitive stimuli, exposure in vivo for avoided movements).
  Stage IV. Maintenance (Identifying key elements, Planning for flare-ups).
  Interventions: Behavioral: Hybrid
- internet Cognitive Behavior Therapy (iCBT) (Active Comparator): CBT pain treatment, delivered via the internet consists of 8, weekly, modules and includes topics such as pain education, pain coping strategies (e.g. pacing), relaxation, cognitive restructuring, problem solving, stress and sleep management, conflict resolution. Patients read materials included in each module and do homework tasks on which they report back to the therapist via the internet. The therapist gives written feedback and guidance after each module. See reference for details.
  Interventions: Behavioral: internet Cognitive Behavior Therapy (iCBT)

INTERVENTIONS:
Behavioral: Hybrid — The hybrid emotion-focused treatment integrates procedures from exposure and dialectical behavior therapy (DBT) with a clear uniting conceptualization focused on targeting underlying processes that maintain co-occurring chronic pain and emotional problems.
  Arms: Hybrid
Behavioral: internet Cognitive Behavior Therapy (iCBT) — A state-of-the-art CBT pain treatment, delivered via the internet.
  Arms: internet Cognitive Behavior Therapy (iCBT)

SUMMARY:
The aim of this project is to evaluate a hybrid emotion-focused treatment protocol, specifically developed for individuals who suffer from co-occurring chronic pain and clinical levels of anxiety and/or depressive symptoms.

Specific questions relating to treatment outcome:

1. Does a hybrid emotion-focused treatment lead to a decrease in comorbid emotional symptoms (pain-related fear, anxiety, depression)?
2. Does a hybrid emotion-focused treatment lead to an increase in functional ability, improvement in work status and decrease in medication use?
3. Does a hybrid emotion-focused treatment lead to better treatment effect on the above outcome variables compared to an active comparison group?

   Specific questions relating to the process of change:
4. Are therapeutic effects of the hybrid emotion-focused treatment mediated by changes in proposed transdiagnostic emotion regulation process variables (worry, rumination, cognitive and behavioral avoidance, emotional suppression)?

DETAILED DESCRIPTION:
Design. A randomized controlled trial in which chronic pain patients with co-occurring emotional problems will receive either:

1. A hybrid individual treatment combining emotion regulation focused Dialectical Behavior Therapy (DBT) with standard exposure methodology. The treatment targets the transdiagnostic psychological processes that have been shown to maintain emotional dysregulation.
2. An active control condition receiving internet-delivered pain management treatment based on Cognitive Behavioral principles. This treatment is evidence-based and thus provides a credible and ethical active comparison group.

Selection. N=84 (ES=.5, p=.05 and ß=.80; based on an estimated between group difference on the Hospital Anxiety and Depression Scale, and compensating for an approximate drop out rate of 20% per condition). Patients will be recruited through pain rehabilitation units in Orebro and Linkoping and via advertisements in the local newspapers.

Procedure. Patients will be examined and screened by trained professionals to exclude individuals with red flags (serious medical illnesses that explain pain conditions), a risk of suicide, and/or need of emergency psychiatric care. After screening and baseline assessment, participants will be randomized to receive either the individual face-to-face hybrid emotion focused treatment (10-15 weekly or biweekly sessions) or the individual, guided, internet-based Cognitive Behavior Therapy (iCBT) treatment for pain (10 weekly sessions). The internet treatment is therapist guided through email contact. The hybrid treatment will be conducted by a trained and supervised licensed clinical psychologist and the internet guidance will be provided by trained and supervised clinical psychologists in their final stage of clinical training. The hybrid emotion-focused treatment integrates procedures from exposure and DBT with a clear uniting conceptualization focused on targeting underlying processes that maintain co-occurring chronic pain and emotional problems.

ELIGIBILITY:
Inclusion Criteria:

* Chronic musculoskeletal pain (> 6 months duration), not emanating from malignancies, systemic diseases (e.g. rheumatoid arthritis) or localized single-joint osteoarthritic conditions in the lower extremities (e.g. knee-osteoarthritis, hip- osteoarthritis).
* Functional problems due to pain (defined as > 10 points on question 21-24 of the Orebro Musculoskeletal Pain Questionnaire).
* Emotional problems (defined as >7 points (cut-off for a probable case) on at least one of the two subscales (anxiety and depression) of the Hospital Anxiety and Depression Scale).

Exclusion Criteria:

* Severe psychiatric disorders that may require immediate other treatment (alcohol abuse, bipolar disorder, psychotic disorders),
* Currently in psychological treatment elsewhere,
* Recently been started on psychopharmacological treatment for depression and/or anxiety (cut off criterion: < 3 months prior to planned treatment start),
* Insufficient mastery of the Swedish language written as well as spoken,
* No personal computer available.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2016-01; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg depression rating scale (MADRS) change | baseline, 3 months, 12 months
  change in self rated depression (from pretreatment, to post treatment and follow up) Scale range 0-60 (higher values worse outcome)
Multidimensional Pain Inventory (MPI) change | baseline, 3 months, 12 months
  change in pain intensity and interference (from pretreatment, to post treatment and follow up). Subscale pain intensity range 0-12, subscale pain interference range 0-66 (for both subscales higher values worse outcome)
Pain Catastrophizing Scale (PCS) change | baseline, 3 months, 12 months
  change in pain catastrophizing (from pretreatment, to post treatment and follow up). Scale range 0-52 (higher values worse outcome).
Generalised Anxiety Disorder 7-item Scale (GAD-7) change | baseline, 3 months, 12 months
  change in general anxiety (from pretreatment, to post treatment and follow up). Scale range 0-27 (higher values worse outcome).

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS) change | baseline, 1.5 months, 3 months
  change in emotion regulation (from pretreatment, to mid- and post treatment)
The Behavior Activation for Depression Scale (BADS) change | baseline, 1.5 months, 3 months
  change in behavioral activation (from pretreatment, to mid- and post treatment)
Self-Compassion scale-12 (SCS) change | baseline, 3 months
  change in self compassion (from pretreatment to post treatment)
Insomnia Severity Index (ISI) change | baseline, 3 months
  change in insomnia (from pretreatment to post treatment)
Tampa Scale for Kinesiophobia (TSK) change | baseline, 3 months
  change in fear avoidance (from pretreatment to post treatment)
Chronic Pain Acceptance Questionnaire (CPAQ) change | baseline, 3 months
  change in pain acceptance (from pretreatment to post treatment)
Lisat 11 change | baseline, 3 months, 12 months
  change in quality of life (from pretreatment to post treatment and follow up)

OTHER OUTCOMES:
adverse effects | 3 months
  adverse treatment effects, measured post treatment
treatment satisfaction questionnaire | 3 months
  self report satisfaction with treatment measured at post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Katja Boersma, PhD, Principal Investigator — Örebro University, Sweden
Locations (2):
- Sweden (2):
  - Smärt- och rehabiliteringscentrum Linköping, Linköping
  - Center for Health and Medical Psychology, Örebro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buhrman M, Nilsson-Ihrfeldt E, Jannert M, Strom L, Andersson G. Guided internet-based cognitive behavioural treatment for chronic back pain reduces pain catastrophizing: a randomized controlled trial. J Rehabil Med. 2011 May;43(6):500-5. doi: 10.2340/16501977-0805. PMID 21533329